CLINICAL TRIAL: NCT03659838
Title: Luftibus in the School: a Population-based Study of Respiratory Symptoms, Lung Function and Air Pollution.
Brief Title: Luftibus in the School: a Study on the Respiratory Health of Schoolchildren.
Acronym: LUIS
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: LUIS
Record Dates: First submitted 2018-07-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Disease
Keywords: Asthma; Wheeze; Cough; Snoring; Bronchial obstruction; Air pollution
MeSH Terms: conditions — Respiration Disorders; Asthma; Respiratory Sounds; Cough; Snoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Schoolchildren from the canton of Zürich aged 6 to 16 years

SUMMARY:
This study assessed the respiratory health of schoolchildren from the canton of Zurich by combining self-reported information on respiratory symptoms with lung function test results and air pollution measurements.

Luftibus in the school (LUIS) is a population-based study conducted in the canton of Zurich, Switzerland. Between the years 2013 and 2016 a bus with equipment for lung function testing and air pollution measurement visited numerous schools across the canton Zurich. The parents of the schoolchildren filled in a questionnaire with validated questions on upper and lower respiratory symptoms, trigger factors, diagnosis, treatment of respiratory symptoms, health behavior and environmental factors. The children were interviewed using a shorter questionnaire. Fieldworkers measured lung function (spirometry and double tracer gas single-breath washout) and an airway inflammation test (fractional exhaled nitric oxide) in the bus. The recruited population included 3500 schoolchildren aged 6 to 16 years from the canton of Zurich.

Respiratory symptoms and their influence on physical activity and sleep have a strong impact on children's quality of life and school performance. The results of this study will provide new insights on schoolchildren's respiratory health that may help to establish new recommendations and influence policy makers' decisions.

DETAILED DESCRIPTION:
Background:

Few population-based studies have recently investigated the epidemiology of childhood respiratory symptoms in Switzerland.

Objectives:

The Luftibus in the school study was setup to assess the respiratory health of schoolchildren from the canton of Zurich and to investigate relationships between respiratory symptoms, lung function and air pollution.

Methods:

Recruitment and participation:

All schools in the canton of Zürich were invited to participate in the LUIS study. Those schools interested in participating were approached. The eligible study population were children aged 6 to 16 years with parental consent from the schools that agreed to participate. Prior to each school visit, parents received a letter with information about the project, an informed consent form and a questionnaire. During the school visit, trained field workers performed lung function tests in children at the school, interviewed the children using a short questionnaire and collected the parental questionnaires. A subsample of the schools was visited again one year after the first visit in order to collect follow-up information, using the same procedure and gathering the same measurements.

Information collected:

- Parental questionnaire: Frequency, duration, severity, triggers of upper and lower respiratory symptoms, previous doctor diagnosis of asthma, use of medication, health behaviors, environmental factors, household characteristics and family history.

- Children's questionnaire: Respiratory symptoms, asthma diagnosis, medication and smoking.

- Anthropometric data: Height and weight were measured by fieldworkers in the schools in a standardized way.

- Complementary tests: Spirometry, fractional exhaled nitric oxide (FeNO) and double tracer gas single-breath washout (SBW) were performed in the school by trained fieldworkers according to ATS criteria.

- Air pollution measurements: Air pollution detectors placed on the roof of the bus measured nitrogen dioxide (NO2), inhalable particles of 10 micrometers or less in diameter (PM10) and ozone concentration at the school site.

Study database:

The study questionnaire database was created using Epidata, which allows data entry and data extraction in CVS format.

Funding:

Lung League of Zurich

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren living in the canton of Zürich
* Age range 6 to 16 years
* Parental consent to participate

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample of schoolchildren from the canton of Zürich
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2013-11-28 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Parent-reported respiratory symptoms | At baseline
  Prevalence of upper and lower respiratory tract symptoms including wheeze, cough, rhinitis and snoring, reported using parent questionnaires.
Self-reported respiratory symptoms | At baseline
  Prevalence of upper and lower respiratory tract symptoms including wheeze, cough, rhinitis and snoring, reported using participant questionnaires.
Lung function measurements: Spirometry, forced expiratory volume in 1 second z-scores | At baseline
  Forced expiratory volume in 1 second (FEV1) z-scores calculated based on Global Lung Function Initiative (GLI) reference values.
Lung function measurements: Spirometry, forced vital capacity z-scores | At baseline
  Forced vital capacity (FVC) z-scores calculated based on Global Lung Function Initiative (GLI) reference values.
Lung function measurements: Single-breath washout | At baseline
  Slope from the tidal (alveolar) phase III (SIII) from double-tracer gas single-breath washout test curves.
Airway inflammation | At baseline
  Airway inflammation measured by levels of fractional concentration of exhaled nitric oxide.

SECONDARY OUTCOMES:
Parent-reported respiratory symptoms | One year after baseline
  Prevalence of upper and lower respiratory tract symptoms including wheeze, cough, rhinitis and snoring, reported using parent questionnaires.
Self-reported respiratory symptoms | One year after baseline
  Prevalence of upper and lower respiratory tract symptoms including wheeze, cough, rhinitis and snoring, reported using participant questionnaires.
Lung function measurements: Spirometry, forced expiratory volume in 1 second z-scores | One year after baseline
  Forced expiratory volume in 1 second (FEV1) z-scores calculated based on Global Lung Function Initiative (GLI) reference values.
Lung function measurements: Spirometry, forced vital capacity z-scores | One year after baseline
  Forced vital capacity (FVC) z-scores calculated based on Global Lung Function Initiative (GLI) reference values.
Lung function measurements: Single-breath washout | One year after baseline
  Slope from the tidal (alveolar) phase III (SIII) from double-tracer gas single-breath washout test curves.
Airway inflammation | One year after baseline
  Airway inflammation measured by levels of fractional concentration of exhaled nitric oxide.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Möller, PD Dr.med, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Researchers wanting to use the Luftibus in the school dataset can contact the study team and propose a research topic. A concept sheet describing the planned analyses and publication must be approved by the Luftibus in the school study team.
  For further details, contact:
  Alexander.Moeller@kispi.uzh.ch Claudia.Kuehni@ispm.unibe.ch

REFERENCES:
- [Derived] Kentgens AC, Kurz JM, Mozun R, Usemann J, Pedersen ESL, Kuehni CE, Latzin P, Moeller A, Singer F; LuftiBus In the School (LUIS) Study Group. Evaluation of the Double-Tracer Gas Single-Breath Washout Test in a Pediatric Field Study. Chest. 2024 Feb;165(2):396-404. doi: 10.1016/j.chest.2023.09.006. Epub 2023 Sep 15. PMID 37716474